CLINICAL TRIAL: NCT00997516
Title: A Randomized, Controlled Trial of Single-incision Laparoscopic (SILS) Versus Conventional Laparoscopic Appendectomy for the Treatment of Acute Appendicitis
Brief Title: Single-incision Laparoscopic (SILS) Versus Conventional Laparoscopic Appendectomy for the Treatment of Acute Appendicitis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Planned interim analysis showed worse outcomes in experimental group
Sponsor: University of California, San Francisco (Other)
Collaborators: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UCSF SILS 01
Record Dates: First submitted 2009-10-15; First posted 2009-10-19 (Estimated); Results first posted 2014-08-22 (Estimated); Last update posted 2014-08-22 (Estimated); Status verified 2014-08

CONDITIONS: Appendicitis
Keywords: Laparoscopy; Appendicitis; Single-incision laparoscopic surgery; SILS
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SILS appendectomy (Experimental): The study population will consist of patients who come to the emergency room with acute abdominal pain and are found to have acute appendicitis on the basis of clinical evaluation and CT of the abdomen/pelvis.
  Interventions: Procedure: SILS appendectomy
- Conventional laparoscopic appendectomy (Active Comparator): The study population will consist of patients who come to the emergency room with acute abdominal pain and are found to have acute appendicitis on the basis of clinical evaluation and CT of the abdomen/pelvis.
  Interventions: Procedure: conventional laparoscopic appendectomy

INTERVENTIONS:
Procedure: SILS appendectomy — Use of SILSPort to perform laparoscopic appendectomy
  Arms: SILS appendectomy
Procedure: conventional laparoscopic appendectomy — conventional laparoscopic removal of the appendix
  Arms: Conventional laparoscopic appendectomy

SUMMARY:
Recent advances in laparoscopic instrumentation have made it possible to perform intra-abdominal operations entirely through a small incision that can be hidden within the umbilicus. The goal is to perform surgery with fewer incisions and no visible scars. Other potential benefits are faster recovery, less pain, and fewer wound complications. The term SILS (Single Incision Laparoscopic Surgery) is being used to describe such techniques, and many have touted SILS as a major breakthrough in minimally-invasive surgery, moving the field closer to surgery that is bloodless, incisionless, and painless. Despite the hype, prospective comparisons of SILS versus conventional laparoscopy are lacking. Results of SILS procedures have generally been limited to case reports and small case series that lack controls. The investigators propose to conduct a prospective, randomized, single-center trial of SILS appendectomy versus conventional laparoscopic appendectomy to treat acute appendicitis. Primary end-points are operative time, complication rate, postoperative pain, recovery time, and long-term cosmetic outcome. The investigators hypothesize SILS appendectomy is equivalent to laparoscopic appendectomy with respect to operative time, complication rate, postoperative pain, and recovery time while providing a better cosmetic outcome.

DETAILED DESCRIPTION:
EXPERIMENTAL DESIGN AND METHODS Patient Enrollment: The study population will consist of patients who come to the emergency room with acute abdominal pain and are found to have acute appendicitis on the basis of clinical evaluation and CT of the abdomen/pelvis. At UCSF, such patients are first evaluated by a small group of general surgeons who provide emergency consultations. Once a decision to operate has been made on clinical grounds, the principal investigator (Dr. Carter) or his delegate will be contacted to approach the patient for enrollment and informed consent.

All patients will receive standard care which consists of preoperative broad-spectrum antibiotics consisting of Zosyn, Ertapenem, or Cipro/Flagyl and intravenous fluids.

Surgeon Enrollment: All surgeons at UCSF who take call in the Emergency Department routinely perform conventional laparoscopic appendectomy for acute appendicitis. Surgeons wishing to participate in the trial will perform 5 proctored SILS appendectomies outside of the trial before enrolling patients. We chose the number 5 because one study showed that SILS operative times (a surrogate for procedural mastery) leveled off by the 5th case for surgeons already proficient in laparoscopy.

Randomization: After enrollment, patients will be assigned to conventional laparoscopic appendectomy versus SILS appendectomy in a 1:1 ratio by a computerized random number generator (http://www.random.org). Even-numbered patients will receive conventional laparoscopic appendectomy, odd-numbered will receive SILS appendectomy.

Conventional laparoscopic appendectomy technique: Patients are placed in the supine position and given a general anesthetic. An orogastric tube is placed. Sequential compression devices are placed on the legs. Unless the patient has just voided, a Foley catheter is placed in the bladder. The left arm is tucked and the abdomen shaved as necessary. The umbilical skin is anesthetized with 5mL of 0.25% marcaine. A 1.5cm vertical or transverse skin incision is made within the umbilical stalk, the fascia is retracted, and a 1.5cm vertical fascial incision made with a scalpel. A 12mm Hasson port is placed through the fascia and the abdomen insufflated to 15mmHg with carbon dioxide gas. Alternatively, a small nick in the fascia can be made, a Veress needle used to achieve pneumoperitoneum, and a 12mm VersSTEP port placed through an introducer sheath. Diagnostic laparoscopy is then performed, with inspection of the stomach, liver, gallbladder, colon, small intestines, and pelvis. If a diagnosis other than acute appendicitis is made (such as pelvic inflammatory disease, sigmoid diverticulitis, cecal diverticulitis, Crohn's disease, perforated duodenal ulcer, etc.), the patient is excluded from the study and treated appropriately. If the appendix looks normal and no other pathology is found in the abdomen, the patient may stay enrolled in the study if the surgeon decides to remove the appendix.

Additional 5mm ports are placed in the left lower quadrant and suprapubic midline after the skin and peritoneum are anesthetized with 0.25% marcaine. A 5mm camera is transferred to the left lower quadrant port site and the appendix is exposed and retracted anteriorly. The mesoappendix may be divided with EndoGIA staplers, Ligasure, cautery and clips, or Harmonic Scalpel. The base of the appendix may be ligated with EndoGIA staplers or Endoloop. The appendix is removed through the umbilical incision after first placing it into an EndoCatch bag. Minimal irrigation is used; perforated cases are treated with suctioning of intra-abdominal pus and postoperative antibiotics. Blood loss is estimated. Umbilical fascia length is measured in millimeters, then closed with 0-Maxon absorbable suture. The umbilical skin is anesthetized with 0.25% marcaine, and all skin edges re-approximated with 4-0 biosyn. Indermil glue is the only dressing.

SILS Appendectomy Technique: Patients are placed in the supine position and given a general anesthetic. An orogastric tube is placed. Sequential compression devices are placed on the legs. Unless the patient has just voided, a Foley catheter is placed in the bladder. The left arm is tucked and the abdomen shaved as necessary. The base of the umbilical stalk is everted by two penetrating towel clamps placed either side of the midline. The skin is anesthetized with 5mL of 0.25% marcaine. A vertical skin incision is made within the umbilical stalk, the fascia is retracted, and a 3 cm vertical fascial incision made with a scalpel. The peritoneum is entered with either a gloved finger, Kelly clamp, or scissors. The incision is retracted anteriorly with an Army/Navy retractor, and the SILSPort inserted into the incision using a shoe-horn maneuver. 5mm trocars are placed in the SILSPort™, and the abdomen insufflated to 15mmHg with carbon dioxide gas, after which the trocars are repositioned into a staggered elevation. Diagnostic laparoscopy is then performed, with inspection of the stomach, liver, gallbladder, colon, small intestines, and pelvis. If a diagnosis other than acute appendicitis is made (such as pelvic inflammatory disease, sigmoid diverticulitis, cecal diverticulitis, Crohn's disease, perforated duodenal ulcer, etc.), the patient is excluded from the study and treated appropriately. If the appendix looks normal and no other pathology is found in the abdomen, the patient may stay enrolled in the study if the surgeon decides to remove the appendix.

The appendix is exposed and retracted anteriorly. The mesoappendix may be divided with EndoGIA staplers, Ligasure, cautery and clips, or Harmonic Scalpel. The base of the appendix may be ligated with EndoGIA staplers or Endoloop. When staplers are used, one of the 5mm trocars is replaced with a 12mm trocar. The appendix is removed through the umbilical incision after first placing it into an EndoCatch bag. Minimal irrigation is used; perforated cases are treated with suctioning of intra-abdominal pus and postoperative antibiotics. Blood loss is estimated. Umbilical fascia length is measured in millimeters, then closed with 0-Maxon absorbable simple interrupted sutures. Skin edges re-approximated with 4-0 biosyn. Indermil glue is the primary dressing.

Postoperative Care: Patients are given a full liquid diet immediately after surgery, and are advanced to an unrestricted diet as soon as the patient feels up to it. Pain is controlled by a hydromorphone PCA (patient-controlled analgesia) pump for at least 12 hours after surgery, after which oral pain medications are prescribed. If the patient is allergic to hydromorphone, morphine may be used. No supplemental pain medications (Motrin, Toradol, etc.) will be used for patients enrolled in the study. No steroids (e.g. Decadron) will be given. Antibiotics for appendicitis are given at the discretion of the attending surgeon. Patients are discharged at the discretion of the attending surgeon, generally when the patient can eat without vomiting, pain is controlled with oral medications, and the systemic inflammatory response to the appendicitis has subsided.

After 2-3 weeks, follow-up occurs in Dr. Carter's clinic. The wounds are assessed for infection, seroma, or hernia. Date of return-to-work and date of last opiate pain medication are recorded. At 6 months, patients return to clinic and complete a survey. The survey includes a Body Image Questionnaire, a Cosmetic Appearance Scale, and a Photo Series Questionnaire, all of which have been validated.8-12 The Body Image Questionnaire measures patients' perception of and satisfaction with their own body and explores attitudes toward their bodily appearance. Five questions are asked, with up to four points assigned per question, totaling 20 possible points. The Cosmetic Appearance Scale assesses the degree of patient satisfaction about the physical appearance of the abdomen (and its scars) using 100-mm visual analogue scale. The patient is asked to make a mark along the horizontal scale that indicates the overall aesthetic appearance of the abdomen as a whole, and incisions separately. Numeric scores are then obtained by measuring the horizontal distance from the low end of the scale to the marking, rounded to the nearest millimeter. Finally, the Photo Series Questionnaire assesses whether knowledge of the cosmetic results of the alternative approach (SILS or conventional laparoscopic) influences the evaluation of the scar. It also measures the strength of the preference. Patients who do not return for follow-up will be mailed a survey and/or called for a telephone interview. Data management and interviews will be managed by a research assistant hired for the study.

Definition of Study Variables and Outcome Measures Patient Characteristics: Age, height, weight, prior operations in the abdomen

Intraoperative Variables:

1. Operative time - defined as the amount of time to perform the operation from skin-incision to application of the dressing. This time is routinely charted by the circulating nurse in the operating room.
2. Conversion - defined by the use of incisions and/or trocars in addition to the ones described in the Methods section, or the need to perform an open procedure.
3. Visceral or vascular injury - defined as injury to the intestines, colon, omentum, vasculature, or pelvic organs during the dissection requiring intervention (suture or stapled repair, use of hemostatic agents).
4. Umbilical fascia incision length (in millimeters).

Postoperative Variables:

1. Mean pain score over 12 hours - Pain is assess by the ward nurse as needed, but at least every four hours, and documented in the patient's chart. Pain is scored on a scale of 0-10, 10 being the most severe pain imaginable. Average pain score for that patient is calculated over the first 12 hours (the time the patient is on a hydromorphone PCA)
2. Hydromorphone use over 12 hours - Total hydromorphone usage (in milligrams) is charted by the floor nurse. The amount used in the first 12 hours after surgery, starting from the time the patient is discharged from the recovery room, is recorded.
3. Length of stay - Number of calendar days the patient is hospitalized.
4. Wound infection - Defined as the need for additional antibiotics, prescribed beyond the perioperative antibiotics given for acute appendicitis, for the purpose or treating a wound cellulitis, or the need to open the wound to drain a wound abscess, within 6 months of surgery.
5. Deep space infection - Defined as the need for reoperation, readmission, or percutaneous drainage of a deep (organ space) infection within 6 months of surgery. All intra-abdominal abscesses are classified as deep space infections.
6. Wound seroma - Defined as an un-inflamed fluid collection under the skin incision > 1cm in diameter identified within 6 months of surgery.
7. Time to return to work - Defined as the number of calendar days between discharge from the hospital and the first day back at work.
8. Date of last opiate pain medication use.
9. Readmission with 30 days.
10. Body Image Score at 6 months
11. Cosmetic Appearance Scale at 6 months.
12. Photo Series Questionnaire at 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Suspected acute appendicitis on clinical and radiographic (CT) grounds

Exclusion Criteria:

1. Phlegmon, mass, peri-appendicecal abscess, or diffuse peritonitis
2. Prior open laparotomy with incision through the umbilicus
3. Body Mass Index > 35
4. Age <18 years
5. Mental illness, dementia, or inability to provide informed consent
6. Chronic pain requiring daily medication (including opiate and NSAIDs)
7. Pregnancy
8. Alternative diagnosis found by diagnostic laparoscopy (post-randomization)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2010-05; Primary Completion 2012-12 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan T. Carter, M.D., Principal Investigator — UCSF Department of Surgery
Locations (2):
- United States (2):
  - UCSF Medical Center, San Francisco, California
  - University of California, San Francisco, San Francisco, California

REFERENCES:
- [Background] Palanivelu C, Rajan PS, Rangarajan M, Parthasarathi R, Senthilnathan P, Praveenraj P. Transumbilical endoscopic appendectomy in humans: on the road to NOTES: a prospective study. J Laparoendosc Adv Surg Tech A. 2008 Aug;18(4):579-82. doi: 10.1089/lap.2007.0174. PMID 18721008
- [Background] Chouillard K FA. Single incision appendectomy for acute appendicitis: a preliminary experience. In: SAGES 2009 Scientific Session, April 22-29, Phoenix, AZ (abstract only); 2009.
- [Background] Kravetz AJ ID, Kia MA. Initial experience in single-port laparoscopic appendectomies. SAGES 2009 Scientific Session, April 22-29, Phoenix, AZ (abstract only)
- [Result] Nguyen NT, Reavis KM, Hinojosa MW, Smith BR, Stamos MJ. A single-port technique for laparoscopic extended stapled appendectomy. Surg Innov. 2009 Mar;16(1):78-81. doi: 10.1177/1553350608330528. Epub 2009 Jan 13. PMID 19141492
- [Result] Edwards C BA. Single incision laparoscopic appendectomy is safe and results in excellent cosmetic outcomes. SAGES 2009 Scientific Session, April 22-29, Phoenix, AZ (abstract only) 2009.
- [Derived] Carter JT, Kaplan JA, Nguyen JN, Lin MY, Rogers SJ, Harris HW. A prospective, randomized controlled trial of single-incision laparoscopic vs conventional 3-port laparoscopic appendectomy for treatment of acute appendicitis. J Am Coll Surg. 2014 May;218(5):950-9. doi: 10.1016/j.jamcollsurg.2013.12.052. Epub 2014 Feb 19. PMID 24684867
- See also: Covidien SILSPort website — http://www.sils.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study population consisted of all patients from May 2010 to November 2012 who presented to the emergency department and were diagnosed with acute appendicitis on the basis of clinical and radiographic evaluation.
Pre-assignment Details: 88 patients were assessed for eligibility. 5 patients were excluded because the study surgeon was unavailable to perform the procedure. 6 patients declined to participate.
Groups:
- SILS Appendectomy: SILS appendectomy: Use of SILS Port to perform laparoscopic appendectomy
Period: Short-term Follow-up (Post Operative)
Arm/Group | SILS Appendectomy | Conventional Laparoscopic Appendectomy
Started | 37 | 38
Completed | 37 | 38
Not Completed | 0 | 0
Period: Long-term Follow-up (After 6 Months)
Arm/Group | SILS Appendectomy | Conventional Laparoscopic Appendectomy
Started | 37 | 38
Completed | 31 | 36
Not Completed | 6 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SILS Appendectomy | Conventional Laparoscopic Appendectomy | Total
Number analyzed (Participants) | 37 | 38 | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 34 (11) | 35 (12) | 34 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 14 | 32
  Male | 19 | 24 | 43
Region of Enrollment [Number; unit: participants]
  United States | 37 | 38 | 75

OUTCOME MEASURES:

1. Primary Outcome: Pain After Surgery
Description: Mean pain score during 12 hours post-surgery, assessed by the ward nurse as needed, but at least every 4 hours, and documented in the patient's chart. Patients were asked to rate their pain on a scale of 0 to 10, with 10 being the most severe pain imaginable and 0 being no pain at all.
Time Frame: 12 hours post-surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SILS Appendectomy | Conventional Laparoscopic Appendectomy
Number analyzed (Participants) | 37 | 38
units on a scale | 4.4 (1.6) | 3.5 (1.5)
Statistical Analysis 1: Comparison: SILS Appendectomy vs Conventional Laparoscopic Appendectomy; Test type: Superiority or Other; p = 0.01, Wilcoxon (Mann-Whitney) — Significant at p<0.05

2. Secondary Outcome: Operative Time
Description: The amount of time to perform the operation from skin-incision to application of the dressing. This time is routinely charted by the circulating nurse in the operating room.
Time Frame: up to 6 hours
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | SILS Appendectomy | Conventional Laparoscopic Appendectomy
Number analyzed (Participants) | 37 | 38
minutes | 54 (17) | 38 (12)
Statistical Analysis 1: Comparison: SILS Appendectomy vs Conventional Laparoscopic Appendectomy; Test type: Superiority or Other; p < 0.01, t-test, 2 sided — Significant at p<0.05

3. Secondary Outcome: Procedures Requiring Conversion to Open or Additional Port
Description: Patients requiring use of additional incisions and/or trocars, or the need to perform an open procedure.
Time Frame: during surgery , up to 6 hours
Measure: Number; unit: participants
Arm/Group | SILS Appendectomy | Conventional Laparoscopic Appendectomy
Number analyzed (Participants) | 37 | 38
participants | 1 | 0

4. Secondary Outcome: Visceral or Vascular Injury
Description: Number of participants who required intervention (suture or stapled repair, use of hemostatic agents) for injury to the intestines, colon, omentum, vasculature, or pelvic organs during the dissection.
Time Frame: during surgery, up to 6 hours
Measure: Number; unit: participants
Arm/Group | SILS Appendectomy | Conventional Laparoscopic Appendectomy
Number analyzed (Participants) | 37 | 38
participants | 0 | 0

5. Secondary Outcome: Length of Stay
Description: Number of calendar days the participant was hospitalized.
Time Frame: up to 14 days
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | SILS Appendectomy | Conventional Laparoscopic Appendectomy
Number analyzed (Participants) | 37 | 38
Days | 1.4 (0.8) | 1.6 (1.8)

6. Secondary Outcome: Wound Infection
Description: Number of participants who required additional antibiotics, prescribed beyond the perioperative antibiotics given for acute appendicitis, for the purpose or treating a wound cellulitis.
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | SILS Appendectomy | Conventional Laparoscopic Appendectomy
Number analyzed (Participants) | 37 | 38
participants | 0 | 0

7. Secondary Outcome: Deep Space Infection
Description: Number of participants who required reoperation, readmission, or percutaneous drainage of a deep (organ space) infection within 6 months of surgery. All intra-abdominal abscesses were classified as deep space infections.
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | SILS Appendectomy | Conventional Laparoscopic Appendectomy
Number analyzed (Participants) | 37 | 38
participants | 1 | 0

8. Secondary Outcome: Wound Seroma
Description: Number of participants who experienced un-inflamed fluid collection under the skin incision > 1cm in diameter identified within 6 months of surgery.
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | SILS Appendectomy | Conventional Laparoscopic Appendectomy
Number analyzed (Participants) | 37 | 38
participants | 1 | 0

9. Secondary Outcome: Time to Return to Work
Description: Number of calendar days between participants' discharge from the hospital and the first day back at work.
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | SILS Appendectomy | Conventional Laparoscopic Appendectomy
Number analyzed (Participants) | 37 | 38
Days | 8.1 (6.2) | 6.9 (4.1)

10. Secondary Outcome: Readmission Within 30 Days.
Description: Number of participants readmitted to the hospital within 30 days of surgery
Time Frame: 30 days
Measure: Number; unit: participants
Arm/Group | SILS Appendectomy | Conventional Laparoscopic Appendectomy
Number analyzed (Participants) | 37 | 38
participants | 2 | 1

11. Secondary Outcome: Body Image Score at 6 Months
Description: After a minimum of 6 months, a Body-Image Questionnaire was sent to participants. The questionnaire has 5 questions, with answers ranging from 1 (Extremely) to 4 (Not at all); lower scores indicate worse satisfaction with and perception of bodily appearance.
  Are you less satisfied with our body since the operation? Do you think the operation has damaged your body? Do you feel less attractive as a results of your operation? Do you feel less feminine or masculine as a result of your operation? Is it difficult to look at yourself naked?
Time Frame: 6 months
Population: 67 of 75 patients completed and returned follow-up surveys
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SILS Appendectomy | Conventional Laparoscopic Appendectomy
Number analyzed (Participants) | 31 | 36
units on a scale
  Overall body satisfaction | 3.5 (1.0) | 3.7 (0.6)
  Damage to body from operation | 3.7 (0.4) | 3.8 (0.4)
  Physical attractiveness affected by operation | 3.8 (0.4) | 4.0 (0.4)
  Femininity/masculinity affected by operation | 4.0 (0.0) | 4.0 (0.2)
  Looking at oneself naked | 3.9 (0.3) | 3.9 (0.2)
Statistical Analysis 1: Comparison: SILS Appendectomy vs Conventional Laparoscopic Appendectomy; Overall body satisfaction; Test type: Superiority or Other; p = 0.86, Wilcoxon (Mann-Whitney) — Significant at p<0.05
Statistical Analysis 2: Comparison: SILS Appendectomy vs Conventional Laparoscopic Appendectomy; Damage to body; Test type: Superiority or Other; p = 0.18, Wilcoxon (Mann-Whitney) — Significant at p<0.05
Statistical Analysis 3: Comparison: SILS Appendectomy vs Conventional Laparoscopic Appendectomy; Physical attractiveness; Test type: Superiority or Other; p = 0.04, Wilcoxon (Mann-Whitney) — Significant at p<0.05
Statistical Analysis 4: Comparison: SILS Appendectomy vs Conventional Laparoscopic Appendectomy; Masculinity/femininity; Test type: Superiority or Other; p = 0.34, Wilcoxon (Mann-Whitney) — Significant at p<0.05
Statistical Analysis 5: Comparison: SILS Appendectomy vs Conventional Laparoscopic Appendectomy; Looking at oneself naked; Test type: Superiority or Other; p = 0.63, Wilcoxon (Mann-Whitney) — Significant at p<0.05

12. Secondary Outcome: Satisfaction With Physical Appearance of Abdomen and Scars at 6 Months.
Description: The Cosmetic Appearance Scale assessed the degree of satisfaction with the physical appearance of the abdomen (and its scars) using a visual analogue scale. Numeric scores were obtained by measuring the horizontal distance from the low end of the scale to the marking, and then normalized on a scale of 0-20 points. Higher scores indicate a higher degree of satisfaction.
  Since your operation, how would you describe the overall appearance of your abdomen? (Revolting; Beautiful) Since your operation, how would you describe your incisional scars? (Revolting; Beautiful) How satisfied are you with your incisional scars? (Very unsatisfied; Very satisfied) How much discomfort do your incisional scars cause? (Severe, daily pain; No pain at all) Can you score your own incisional scar? (Worst possible scar; Best possible scar)
Time Frame: 6 months
Population: Participants who returned surveys for long-term follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SILS Appendectomy | Conventional Laparoscopic Appendectomy
Number analyzed (Participants) | 31 | 36
units on a scale
  Appearance of abdomen | 16.3 (3.5) | 15.4 (3.7)
  Appearance of scars | 16.5 (3.2) | 14.4 (4.1)
  Satisfaction with scars | 18.5 (2.2) | 16.9 (3.7)
  Discomfort of scars | 18.6 (2.9) | 18.6 (2.4)
  Overall impression of scars | 18.4 (2.7) | 16.4 (3.0)
Statistical Analysis 1: Comparison: SILS Appendectomy vs Conventional Laparoscopic Appendectomy; Cosmetic appearance of abdomen; Test type: Superiority or Other; p = 0.48, t-test, 2 sided — Significant at p<0.05
Statistical Analysis 2: Comparison: SILS Appendectomy vs Conventional Laparoscopic Appendectomy; Cosmetic appearance of scars; Test type: Superiority or Other; p = 0.09, t-test, 2 sided — Significant at p<0.05
Statistical Analysis 3: Comparison: SILS Appendectomy vs Conventional Laparoscopic Appendectomy; Satisfaction with scars; Test type: Superiority or Other; p = 0.25, t-test, 2 sided — Significant at p<0.05
Statistical Analysis 4: Comparison: SILS Appendectomy vs Conventional Laparoscopic Appendectomy; Discomfort of scars; Test type: Superiority or Other; p = 0.81, t-test, 2 sided — Significant at p<0.05
Statistical Analysis 5: Comparison: SILS Appendectomy vs Conventional Laparoscopic Appendectomy; Overall impression of scars; Test type: Superiority or Other; p < 0.01, t-test, 2 sided — Significant at p<0.05

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | SILS Appendectomy | Conventional Laparoscopic Appendectomy
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/38
Other Adverse Events (participants affected / at risk) | 5/37 | 4/38
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SILS Appendectomy (N=37) | Conventional Laparoscopic Appendectomy (N=38)
Deep space infection (Infections and infestations) | 1 | 0 — Reoperation, readmission, or percutaneous drainage of a deep (organ space) infection within 6 months of surgery
Wound seroma (Skin and subcutaneous tissue disorders) | 1 | 0 — Un-inflamed fluid collection under the skin incision, >1cm in diameter, identified within 6 months of surgery
Postoperative bleeding (Injury, poisoning and procedural complications) | 0 | 1
Urinary retention (Renal and urinary disorders) | 2 | 2
Prolonged postoperative ileus (Gastrointestinal disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes